CLINICAL TRIAL: NCT07358598
Title: The Relationship Between Eye Movement Parameters and Cognitive Functions in Older Adults
Brief Title: Eye Movement Parameters and Cognitive Functions in Older Adults
Status: Not yet recruiting | Type: Observational
Sponsor: National Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: KSVGH24-CT10-11
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Dysfunction
Keywords: Eye movements; Cognitive function impairment; Older adults
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy group-patients with intact cognitive function
- Mild cognitive impairment group-patients with mild cognitive impairment
- Dementia group-patients with severe cognitive impairment

SUMMARY:
Dementia most commonly occurs in elderly individuals, but currently there is still a lack of objective measurement methods that can detect cognitive impairment in older adults at an early stage. Eye movement is considered a clinical indicator with potential for screening mild cognitive dysfunction, and eye movement signals can be extracted to objectively evaluate cognition. Eye tracking has been used mostly to evaluate patients with neurodegenerative diseases such as Parkinson's disease. However, less attention has been paid to the relationship between eye movement and cognitive function in elderly individuals, as well as the association between eye movement data and abnormal cognitive subdomains. This cross-sectional study will recruit 0204 elderly individuals over the age of 65, divided into three groups (healthy group/mild cognitive impairment group/dementia group) according to the purpose of this study. Participants who have not been diagnosed with neurological diseases (such as Parkinson's disease or stroke), or have mental illness or visual impairments will be excluded. This study hopes to provide empirical data on eye movement signals and cognitive function in healthy older individuals, as well as to serve as a preliminary study for future development of eye activity stimulation to improve cognitive function in older adults.

ELIGIBILITY:
Inclusion Criteria:

- Participants are aged 65 years or older and have completed a comprehensive geriatric assessment (CGA) in the outpatient clinic.

Exclusion Criteria:

* Participants are under 65 years of age or those who ar are unable to comply with study procedures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: A total of 210 participants will be recruited, with an estimated 70 individuals in each cognitive group.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2026-01-17 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Eye-tracking measurement | A single assessment is conducted at one study visit (cross-sectional design).
  Eye movement behavior will be assessed as an objective measure of cognitive control in older adults. Eye-tracking data will be collected using the J7EF Gaze Smart Glasses (Jorjin Technologies), a non-invasive wearable eye-tracking system with a sampling frequency of 30 Hz. Participants will perform standardized visual tasks while eye movement behavior is recorded.
  Outcome measures will include task-related eye movement patterns, such as gaze behavior and saccadic performance, which reflect attentional control and higher-order cognitive processing. Alterations in these eye movement parameters have been associated with cognitive impairment. Eye movement measures will be used to characterize differences in cognitive function across participant groups.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | A single assessment is conducted at one study visit (cross-sectional design).
  The Mini-Mental State Examination (MMSE) is a widely used cognitive screening tool originally developed by Folstein and McHugh in 1975 (Folstein et al., 1975). It consists of 30 items assessing six domains of cognitive function: orientation, attention, memory, language, verbal comprehension, praxis, and constructional ability. Higher scores indicate better cognitive function. A total score between 24 and 30 suggests intact cognitive function; scores between 18 and 23 are indicative of mild cognitive impairment; and scores from 0 to 17 reflect moderate to severe cognitive impairment.
  In the present study, the MMSE is used to classify adults aged 65 years and older into cognitive status groups, including a cognitively healthy group, a mild cognitive impairment (MCI) group, and a dementia group, based on established score thresholds.

OTHER OUTCOMES:
Eye-Tracking Task 1: Horizontal Fixation Task (HFT) | A single assessment is conducted at one study visit (cross-sectional design).
  The FXS task is designed to measure fixation stability. Participants are instructed to fixate on a white dot, that appears sequentially at different screen locations: initially in the center, then alternately to the left and right sides of the screen.Each position is maintained for 5 seconds, during which participants are instructed to maintain their gaze on the white dot. The sequence proceeds as follows: Center (5 seconds), right side (5 seconds), left side (5 seconds), and return to center (5 seconds). The task duration is approximately 20 seconds.
Eye-Tracking Task 2: Vertical Fixation Task (VFT) | A single assessment is conducted at one study visit (cross-sectional design).
  The Vertical Fixation Task is designed to assess vertical saccadic eye movements and fixation stability. A white fixation dot is sequentially displayed on a black background at specific vertical locations. The target is presented at the center of the screen and then alternates between upper and lower positions at 5-second intervals (center-upper-lower-center), with a total task duration of approximately 20 seconds.
Eye-tracking Task 3: Horizontal Pursuit Task (HPT) | A single assessment is conducted at one study visit (cross-sectional design).
  The HPT is designed to evaluate participants' ability to perform smooth horizontal pursuit eye movements. A white dot then appears at the center of a black screen, prompting participants to fixate and track the dot continuously as it begins moving horizontally. The stimulus moves smoothly and repeatedly from left to right and back across the screen. Participants are instructed to visually follow the moving dot toward to left and right side without shifting their head position. The task duration is approximately 30 seconds.
Eye-Tracking Task 4: Vertical Pursuit Task (VPT) | A single assessment is conducted at one study visit (cross-sectional design).
  The VPT is designed to evaluate participants' ability to perform smooth horizontal pursuit eye movements. A white dot then appears at the center of a black screen, prompting participants to fixate and track the dot continuously as it begins moving vertically. The stimulus moves smoothly and repeatedly from up to down across the screen. Participants are instructed to visually follow the moving dot toward to up and down side without shifting their head position. The task duration is approximately 30 seconds.
Eye-Tracking Task 5: Horizontal Saccade Task (HST) | A single assessment is conducted at one study visit (cross-sectional design).
  The HST is designed to evaluate rapid, reflexive saccadic eye movements in response to abrupt horizontal target shifts. A white fixation dot appears at the center of the screen and then jumps alternately between the far left and far right positions. Participants are instructed to track the dot continuously from left to right for the entire duration of the task (approximately 30 seconds). Each positional shift is abrupt, requiring quick and accurate horizontal saccades.
Eye-Tracking Task 6: Vertical Saccade Task (VST) | A single assessment is conducted at one study visit (cross-sectional design).
  The VST is designed to evaluate rapid, reflexive saccadic eye movements in response to abrupt horizontal target shifts. A white fixation dot appears at the center of the screen and then jumps alternately between the far up and far down positions. Participants are instructed to track the dot continuously from up to down for the entire duration of the task (approximately 30 seconds). Each positional shift is abrupt, requiring quick and accurate horizontal saccades.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pereira ML, Camargo Mv, Aprahamian I, Forlenza OV. Eye movement analysis and cognitive processing: detecting indicators of conversion to Alzheimer's disease. Neuropsychiatr Dis Treat. 2014 Jul 9;10:1273-85. doi: 10.2147/NDT.S55371. eCollection 2014. PMID 25031536